CLINICAL TRIAL: NCT02630745
Title: Evaluation of the Effect of Immediate and Delayed Surgical Periodontal Therapy After Non-surgical Endodontic Treatment on Periodontal Healing in Concurrent Endodontic Periodontal Lesion With Communication-A Randomized Clinical Trial"
Brief Title: Immediate Verses Delayed Surgical Periodontal Therapy After Endodontic Treatment in Endo Perio Lesion With Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Perio 2
Record Dates: First submitted 2015-12-08; First posted 2015-12-15 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2015-12

CONDITIONS: Attachment Loss; Tooth,Non Vital
Keywords: endodontic treatment; open flap debridement

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate periodontal surgery (Group 1) (Active Comparator): periodontal surgical procedure in the form of open flap debridement will be performed immediately( in which after debridement mucoperiosteal flaps will be repositioned and secured by using 3-0 non-absorbable black silk surgical suture) after obturation of the root canal system( using calcium hydroxide intracanal medicament placed with the help of 27 gauge endodontic syringe for 10 days and access cavity will be sealed with suitable sealer).
  Interventions: Procedure: Immediate periodontal surgery
- Delayed periodontal surgery (Group 2) (Active Comparator): periodontal surgical procedure in the form of open flap debridement( in which after debridement mucoperiosteal flaps will be repositioned and secured by using 3-0 non-absorbable black silk surgical suture) will be performed 3 months after obturation of the root canal system ( using calcium hydroxide intracanal medicament placed with the help of 27 gauge endodontic syringe for 10 days and access cavity will be sealed with suitable sealer).
  Interventions: Procedure: Delayed periodontal surgery

INTERVENTIONS:
Procedure: Immediate periodontal surgery — Treatment involves immediate surgical periodontal therapy in form of open flap debridement after non surgical endodontic treatment and obturation with gutta-percha and zinc oxide eugenol (ZOE) sealer. in concurrent endodontic periodontal lesions with communication .
  Arms: Immediate periodontal surgery (Group 1)
Procedure: Delayed periodontal surgery — Treatment involves surgical periodontal therapy after 3 months of non surgical endodontic treatment and obturation with gutta-percha and zinc oxide eugenol (ZOE) sealer. in the form of open flap debridement in concurrent endodontic periodontal lesions with communication .
  Arms: Delayed periodontal surgery (Group 2)

SUMMARY:
The aim of the study is to conduct a prospective randomized clinical trial to evaluate the effect of immediate and delayed surgical periodontal therapy after non-surgical endodontic treatment on periodontal healing of the concurrent endodontic -periodontal lesion with communication.

DETAILED DESCRIPTION:
Observations based upon review articles and case reports has suggested, if the root canal system is infected, endodontic treatment should be commenced prior to any periodontal therapy in order to remove the intra canal infection before any cementum is removed in case of concurrent endodontic-periodontic lesions without communication. This avoids several complications and provides a more favourable environment for periodontal repair. Treatment results of endodontic therapy should be evaluated in 2-3 months and only then periodontal treatment should be considered. But review articles states that teeth that have concurrent endodontic and periodontal diseases that communicate with each other will require comprehensive treatment with both endodontic and periodontal management. Ideally both infections should be removed before the root canal filling and any final restorations are provided. Completion of the root canal filling should be delayed until the periodontal prognosis has been reassessed and determined following initial, and often further, periodontal treatment. Though Infected root canal systems and periodontal pockets have similar microbiological flora, there are more microbes and more species of spirochetes in periodontal pockets than in infected root canal systems, and the microflora in infected root canals of teeth that have concurrent endodontic and periodontal diseases is more complex than in teeth with infection confined to the periapical region. So the outcome of endodontic treatment may be affected if the root canal filling is placed while there is still a periodontal infection present that communicates with the root canal system since cross-seeding through the apical or lateral foramina is possible. An In-vitro study on human extracted teeth states that despite thorough cleaning and disinfection of the root canal system during endodontic treatment, bacteria from the periodontal lesion may re-invade the root canal system since root canal fillings do not seal canals completely.

All the above findings are based on microbiological,histological,case-reports,retrospective and in-vitro studies.The timing of periodontal treatment in concurrent endodontic -periodontal lesions with communication still remains a issue of debate.No prospective human clinical trial(randomized) has been conducted till date to ascertain whether surgical periodontal treatment should be given immediately after completion of non-surgical endodontic treatment or 2-3 months after completion of non-surgical endodontic treatment.

Thus the aim of our study is to conduct a prospective randomized clinical trial to evaluate the effect of immediate and delayed surgical periodontal therapy after non-surgical endodontic treatment for the management of concurrent endodontic -periodontal lesion with communication.

MATERIAL AND METHOD This randomized clinical trial will be conducted in Department of Periodontics and Oral Implantology in collaboration with Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences, Rohtak.

STUDY POPULATION Patients were recruited from regular out patient department of the department of periodontics and oral implantology,department of conservative dentistry and endodontics and department of oral medicine, diagnosis and radiology. The study will be conducted as follows:-

1. Immediate surgery group Treatment involves surgical periodontal therapy in form of open flap debridement immediately after non-surgical endodontic treatment.
2. Delayed surgery group Treatment involves surgical periodontal therapy in form of open flap debridement 3 months after completion of non-surgical endodontic treatment. INCLUSION CRITERIA Patients of age 18 years and above with a clinical and radiographic diagnosis of combined endodontic periodontal lesion and having generalized chronic periodontitis with at least one non vital tooth having apical radiolucency with communication.

   * Wide base pocket, deep pocket depth
   * Non vital tooth (confirmed by heat test, cold test and electronic pulp test)
   * Radiographic periapical alveolar bone destruction with apical communication
   * Patients having generalized chronic periodontitis [≥2 interproximal sites with clinical attachment level (CAL) ≥ 4mm,not on same tooth(moderate) or ≥2 interproximal sites with clinical attachment level (CAL)≥6mm ,not on same tooth (severe)]26

EXCLUSION CRITERIA

* Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Pregnant or lactating mothers.
* Smokers and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Fractured/perforated roots.
* Developing permanent tooth.
* Previously root canal filled.
* History of recent periodontal treatment within 6 months prior to study.

Prior informed consent will be taken from each patient after explaining the procedure in patient's language along with risk and benefits involved.

METHODOLOGY Patients were randomly allocated to group1 and group 2. The study will be conducted as follows:-

1. Presurgical therapy:- which will be including

   * Oral hygiene instructions
   * Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler, hand scaler and curettes.
   * Conventional root canal therapy will be initiated in both the groups before definite periodontal surgical therapy.
2. Surgical therapy:- In group 1 periodontal surgical procedure in the form of open flap debridement will be performed immediately after obturation of the root canal system In group 2 periodontal surgical procedure in the form of open flap debridement will be performed 3 months after obturation of the root canal system Prior to surgery, a probing stent will be fabricated for every patient,relative to which attachment loss will be measured.

CLINICAL PARAMETERS

1. Full mouth indices to be recorded at baseline

   * Bleeding on probing
   * Probing Pocket depth
   * Attachment loss
2. Site specific indices

   * Plaque index
   * Gingival index
   * Relative Probing Pocket depth
   * Relative attachment loss
   * Bleeding on probing
   * Tooth mobility
   * Relative gingival marginal level Using periodontal probe at 6 sites (mesial, distal, median points at buccal and lingual aspects) per tooth.

Customized bite blocks and parallel angle technique will be used to obtain radiographs Clinical parameters will be recorded at baseline, 3 months and 6 months for Group 1(immediate surgery) Clinical parameters will be recorded at baseline, 3 months, 6 months and 9 months for Group 2(delayed surgery) PERIODONTAL PROCEDURE This involves supragingival and subgingival scaling and root planning to be performed with ultrasonic scaler, hand scaler and curette and will be completed in minimum two sessions.

CONVENTIONAL ENDODONTIC PROCEDURE After achieving local anaesthesia, access opening will be made with the help of round bur. Then the root canal will be thoroughly debrided followed by copious irrigation and subsequently prepared with the help of endo files. After preparation of the canal, calcium hydroxide intracanal medicament will be placed with the help of 27 gauge endodontic syringe for 10 days and access cavity will be sealed with suitable sealer. Obturation will be performed with gutta percha and zinc oxide eugenol based sealer.

PERIODONTAL SURGICAL PROCEDURE After administration of local anaesthesia, buccal and lingual/palatal intracrevicular incision will be made and mucoperiosteal flaps will be reflected including atleast one tooth ahead and another behind the tooth. Meticulous defect debridement and root planning will be carried out using area specific curettes and scalers with special effort to remove all the granulation tissue. After instrumentation, the root surfaces will be washed with saline solution in attempt to remove any remaining detached fragments from the defect and surgical field. After debridement mucoperiosteal flaps will be repositioned and secured by using 3-0 non-absorbable black silk surgical suture. The surgical area will be protected and covered with periodontal dressing and post operative instructions will be given.

Processing of Data Data recorded will be processed by standard statistical analysis.

ELIGIBILITY:
Inclusion Criteria: Patients of age 18 years and above with a clinical and radiographic diagnosis of combined endodontic periodontal lesion and having generalized chronic periodontitis with at least one non vital tooth having apical radiolucency with communication.

* Wide base pocket, deep pocket depth
* Non vital tooth (confirmed by heat test, cold test and electronic pulp test)
* Radiographic periapical alveolar bone destruction with apical communication

Exclusion Criteria:• Systemic illness known to affect the periodontium or outcome of periodontal therapy.

* Patient taking medications such as corticosteroids or calcium channel blockers, which are known to interfere periodontal wound healing or patient on long term NSAID therapy.
* Patients allergic to medication (local anaesthetic, antibiotics, NSAID).
* Pregnant or lactating mothers.
* Smokers and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Fractured/perforated roots.
* Developing permanent tooth.
* Previously root canal filled.
* History of recent periodontal treatment within 6 months prior to study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Relative Attachment Loss | 6 months in group 1, 9 months in group 2
  measurement done by periodontal probe with stents